CLINICAL TRIAL: NCT06794151
Title: Endoscopic Rubber Band Ligation and Milligan-Morgan Hemorrhoidectomy for the Treatment of Grade II-III Internal Hemorrhoids: a Multicenter, Non-randomized Controlled Study
Status: Active, not recruiting | Type: Observational
Sponsor: Weidong Tong (Other)
Responsible Party: Sponsor-Investigator, Weidong Tong, Endoscopic Rubber Band Ligation and Milligan-Morgan Hemorrhoidectomy for the Treatment of Grade II-III Internal Hemorrhoids: A Multicenter, Non-randomized Controlled Study, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: 20241226
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Hemorrhoid
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study adopted a multicenter, non-randomized controlled clinical research design. Patients with internal hemorrhoids who met the inclusion criteria were assigned to the endoscopic rubber band ligation group (observation group) or the Milligan-Morgan hemorrhoidectomy group (control group) according to their treatment preferences. Doctors who were unaware of the clinical data information evaluated the patients' postoperative recovery, the occurrence of complications, and the long-term follow-up of treatment efficacy through outpatient reexaminations, WeChat video calls, or telephone calls.

Research Subjects and Inclusion/Exclusion Criteria 1.1 Research Subjects Patients with grade II-III internal hemorrhoids 1.2 Inclusion Criteria

1. Patients diagnosed with grade II-III internal hemorrhoids according to the Goligher classification;
2. Aged between 18 and 80 years old, both males and females;
3. Those who did not respond well to conservative treatments such as dietary adjustments and medications;
4. Patients who signed the informed consent form and were willing to cooperate with this study.

1.3 Exclusion Criteria

1. Patients with contraindications to colonoscopy;
2. Patients with concurrent anorectal diseases such as anal fissure, anal fistula, thrombosed hemorrhoids, perianal abscess, etc., or a history of previous anorectal surgery;
3. Pregnant patients;
4. Patients with concurrent intestinal infections, inflammatory bowel diseases, or colorectal malignancies;
5. Patients with severe heart, liver, or kidney diseases and coagulation disorders;
6. Patients with diabetes mellitus and poor blood glucose control;
7. Patients with missing clinical data, poor follow-up compliance, or those suffering from mental illnesses and communication disorders;
8. Patients who refused to participate in the study. 1.4 Observation Indicators Primary Indicator: Efficacy Rate Secondary Indicators: Pain, a feeling of fullness and discomfort in the anus, urinary retention, defecation status, long-term therapeutic effect, treatment cost, etc.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients diagnosed with grade II-III internal hemorrhoids according to the Goligher classification; (2) Aged between 18 and 80 years old, both males and females; (3) Those who did not respond well to conservative treatments such as dietary adjustments and medications; (4) Patients who signed the informed consent form and were willing to cooperate with this study.

Exclusion Criteria:

* (1) Patients with contraindications to colonoscopy; (2) Patients with concurrent anorectal diseases such as anal fissure, anal fistula, thrombosed hemorrhoids, perianal abscess, etc., or a history of previous anorectal surgery; (3) Pregnant patients; (4) Patients with concurrent intestinal infections, inflammatory bowel diseases, or colorectal malignancies; (5) Patients with severe heart, liver, or kidney diseases and coagulation disorders; (6) Patients with diabetes mellitus and poor blood glucose control; (7) Patients with missing clinical data, poor follow-up compliance, or those suffering from mental illnesses and communication disorders; (8) Patients who refused to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with grade II-III internal hemorrhoids
Sampling Method: Probability Sample
Enrollment: 548 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy Rate | 6 months
  The primary endpoint of this study is to evaluate the therapeutic effect of hemorrhoids in patients through physical examinations, digital rectal examinations and other means by doctors who are unaware of the clinical data information six months after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, China, Chongqin, China